CLINICAL TRIAL: NCT05862883
Title: Studying the Efficiency of the Natural Preparation Rutan in Children in the Treatment of COVID-19, Acute Respiratory Viral Infections, and Developing Treatment Protocols
Brief Title: Studying the Efficiency of the Natural Preparation Rutan in Children in the Treatment of COVID-19, ARVI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Research Institute of Virology, Ministry of Health of the Republic of Uzbekistan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: А - СС - 2021 - 305
Record Dates: First submitted 2023-05-15; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: COVID-19 Respiratory Infection
Keywords: COVID-19; Rutan; clinical course; laboratory values; effectiveness
MeSH Terms: conditions — COVID-19; Disease Progression | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Main group consisting of 201 children of 6-18 years old with mild and moderate COVID-19 form who were treated at the specialized clinic "Zangiota 1" and were taking Rutan. Control group consisting of 100 children of 6-18 years old with mild and moderate COVID-19 form who were treated at the specialized clinic "Zangiota 1" and were not taking Rutan.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Target group (Experimental): 201 children 6-18 years old with mild to moderate COVID-19, who were taking Rutan.
  Interventions: Drug: Rutan 25 mg
- control group (Other): 100 children 6-18 years old with mild to moderate COVID-19, who were not taking Rutan.
  Interventions: Other: Control group

INTERVENTIONS:
Drug: Rutan 25 mg — Active ingredient: (3,6-bis-O-galloyl-1,2,4-tri-O-galloyl-β-D-glucose). Active substance: "Rutan 25 mg. Excipients: potato starch, calcium stearate, lactulose.
  Other Names: Rutan
  Arms: Target group
Other: Control group — Taking basic therapy without Rutan
  Arms: control group

SUMMARY:
Clinical research includes Determination of efficacy and acceptability of the local medicine "Rutan tablets 0,025" in children and teenagers 6-18 years old with COVID-19 and/or acute respiratory viral infections. And also the purpose of the study was to study clinical and laboratory changes when using Rutan in patients with Covid 19 clinical methods such as collection of anamnesis, dynamic examination of patients, catamnestic observation - a telephone survey, as well as biochemical, immunological, virologic PCR and ELISA tests.

DETAILED DESCRIPTION:
This study is a randomized, open-label, controlled trial to evaluate the safety and efficacy of a novel therapeutic agent, Rutan 25 mg, in hospitalized child patients diagnosed with COVID-19. The study will be a series of comparisons with two groups. The main group will receive the drug "Rutan 25 mg". The control group will not be given the study drug. There will be continuous monitoring to stop the study due to futility, efficacy or safety. Because of the likelihood that the baseline standards for maintenance therapy may evolve/improve over time, safety and efficacy comparisons will adapt.

Randomization will be based on: Card system (the patient will be asked to choose one of two cards with the same drawings on the visible side, and after choosing, when turning over the cards, it will be determined which group the patient will be included) Patients of the main group (210 patients) will be prescribed Rutan 25 mg tablets, along with the therapy recommended at the time of the study. The course of treatment will be - on the first day, 1 tablet 2 times a day. The duration of the course of treatment is 10 days, with good tolerability of the drug.

The comparison group (100 patients) will receive the current recommended treatment at the time of the study without the use of investigational medicine.

Screening failures are defined by participants who agreed to participate in a clinical trial but were not subsequently randomized to participate in the study. A minimum set of information about monitoring failures is required to ensure transparent reporting, compliance with the publication of the Consolidated Reporting Standards (CONSORT), and responses to regulatory requests. The minimum information includes demographics, monitoring failure details, eligibility criteria, and any serious adverse events (SAEs).

Discontinuation of participation/withdrawal of a participant means termination of participation in the study, and the remaining study procedures must be interrupted and replaced by another participant, as indicated in the study protocol. Any clinically significant changes in the patient's condition and/or laboratory values will be reported as an adverse event (AE) by the investigator. The researcher has the right to make changes or terminate the study.

ELIGIBILITY:
Inclusion Criteria:

Submission of a signed and dated informed consent form (guardian). Declared willingness to comply with all study procedures and accessibility during the study.

Children from 6 to 18 years old. Patients with PCR-confirmed COVID-19 with mild/moderate disease. U07.1. Ability to take oral medications and willingness to adhere to the regimen.

Exclusion Criteria:

Severe form of COVID-19. U07.1. Treatment with another investigational drug. Individual intolerance to the drug. The occurrence of any allergic reactions. Weighting of the general well-being of the patient and the transition to a severe form of the disease.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 301 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Effectivness of therapy | twice a day for 10 days
  To evaluate the effectiveness of therapy, a PCR study will be carried out. To determine the severity of the inflammatory syndrome, CRP (C-reactive protein), procalcitonin, ferritin, IL-6, general laboratory tests and general clinical indicators will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Erkin Musabaev, professor, Study Director — +998901869164
Locations (1):
- Tashkent Institute of Virology, Tashkent, Uzbekistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keni R, Alexander A, Nayak PG, Mudgal J, Nandakumar K. COVID-19: Emergence, Spread, Possible Treatments, and Global Burden. Front Public Health. 2020 May 28;8:216. doi: 10.3389/fpubh.2020.00216. eCollection 2020. PMID 32574299
- [Background] Tang T, Bidon M, Jaimes JA, Whittaker GR, Daniel S. Coronavirus membrane fusion mechanism offers a potential target for antiviral development. Antiviral Res. 2020 Jun;178:104792. doi: 10.1016/j.antiviral.2020.104792. Epub 2020 Apr 6. PMID 32272173
- [Background] Gordon DE, Jang GM, Bouhaddou M, Xu J, Obernier K, White KM, O'Meara MJ, Rezelj VV, Guo JZ, Swaney DL, Tummino TA, Huttenhain R, Kaake RM, Richards AL, Tutuncuoglu B, Foussard H, Batra J, Haas K, Modak M, Kim M, Haas P, Polacco BJ, Braberg H, Fabius JM, Eckhardt M, Soucheray M, Bennett MJ, Cakir M, McGregor MJ, Li Q, Meyer B, Roesch F, Vallet T, Mac Kain A, Miorin L, Moreno E, Naing ZZC, Zhou Y, Peng S, Shi Y, Zhang Z, Shen W, Kirby IT, Melnyk JE, Chorba JS, Lou K, Dai SA, Barrio-Hernandez I, Memon D, Hernandez-Armenta C, Lyu J, Mathy CJP, Perica T, Pilla KB, Ganesan SJ, Saltzberg DJ, Rakesh R, Liu X, Rosenthal SB, Calviello L, Venkataramanan S, Liboy-Lugo J, Lin Y, Huang XP, Liu Y, Wankowicz SA, Bohn M, Safari M, Ugur FS, Koh C, Savar NS, Tran QD, Shengjuler D, Fletcher SJ, O'Neal MC, Cai Y, Chang JCJ, Broadhurst DJ, Klippsten S, Sharp PP, Wenzell NA, Kuzuoglu-Ozturk D, Wang HY, Trenker R, Young JM, Cavero DA, Hiatt J, Roth TL, Rathore U, Subramanian A, Noack J, Hubert M, Stroud RM, Frankel AD, Rosenberg OS, Verba KA, Agard DA, Ott M, Emerman M, Jura N, von Zastrow M, Verdin E, Ashworth A, Schwartz O, d'Enfert C, Mukherjee S, Jacobson M, Malik HS, Fujimori DG, Ideker T, Craik CS, Floor SN, Fraser JS, Gross JD, Sali A, Roth BL, Ruggero D, Taunton J, Kortemme T, Beltrao P, Vignuzzi M, Garcia-Sastre A, Shokat KM, Shoichet BK, Krogan NJ. A SARS-CoV-2 protein interaction map reveals targets for drug repurposing. Nature. 2020 Jul;583(7816):459-468. doi: 10.1038/s41586-020-2286-9. Epub 2020 Apr 30. PMID 32353859
- [Derived] Salikhov SI, Abdurakhmonov IY, Oshchepkova YI, Ziyavitdinov JF, Berdiev NS, Aisa HA, Shen J, Xu Y, Xu HE, Jiang X, Zhang L, Vypova NL, Allaberganov DS, Tagayalieva NA, Musabaev EI, Ibadova GA, Rajabov IB, Lokteva LM. Repurposing of Rutan showed effective treatment for COVID-19 disease. Front Med (Lausanne). 2023 Nov 29;10:1310129. doi: 10.3389/fmed.2023.1310129. eCollection 2023. PMID 38093975